CLINICAL TRIAL: NCT00963586
Title: Quality of Life in Patients Treated for Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: University Medical Center Groningen (Other)
Other Study IDs: qol hn maastro umcg
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HNC Maastricht: Patients treated for HNC in the University Hospital Maastricht/MAASTRO clinic, the Netherlands
- HNC Groningen: Patients treated for HNC in the University Medical Center Groningen, the Netherlands

SUMMARY:
Rationale: Due to advanced technologies in the last decade, increasingly more treatment options are available for head and neck cancer (HNC). As a consequence decision-making with regard to choosing the best available treatment option is becoming increasingly relevant. Quality of life weights (utility scores) are an important outcome measure in this decision-making process. Utility scores can be combined with life expectancy, resulting in the Quality Adjusted Life Year (QALY). If in economic evaluation the outcomes are expressed in QALYs gained, it is possible to compare the efficiency of different interventions for different indications. However, limited evidence on utility scores after treatment for HNC is available.

Objective: The investigators' main objective is to examine quality of life (QoL), both utility scores and disease specific quality of life, for different treatment modalities in HNC. Secondary objectives are to examine whether QoL differs across health states, and which factors influence QoL. As extensive data are available on disease-specific quality of life, another objective is to examine whether utility scores can be derived from a commonly used disease-specific questionnaire, the EORTC QLQ-C30/QLQ-H&N35. If this would be possible, this would limit patient burden in future clinical trials. Finally, by means of measuring patients' ability to perform their work, diet and dental consequences the investigators aim to measure the impact of HNC and its treatment.

Study design: The investigators' study design is a cross-sectional survey.

Study population: The study population consists of patients with HNC who are treated at least six months ago for curative radiotherapy and/or surgery with or without chemotherapy.

Intervention/method: Patients are asked to fill out a single set of questionnaires (once-only). The set of questionnaires consists of three validated questionnaires, concerning health state utility (EuroQol-5D), disease-specific quality of life (EORTC QLQ-C30/QLQ-H&N35) and productivity losses (PRODISQ). In addition, two questions inquiring about patients' diet and three questions considering the dental status of these patients are added to the questionnaires. To classify patients into certain health states, physicians are asked to score adverse events in patients during follow-up visits (according to the RTOG classification).

Main study parameters/endpoints: The main study parameter is QoL (both disease specific quality of life and utility scores) in a certain health state. These utility scores can be used in future cost-effectiveness studies to identify the best available treatment option. Other important study parameters are the factors influencing QoL, and the relationship between utility score and disease-specific quality of life.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: As the study involves a once only set of questionnaires, the burden is only minimal. No risks are expected to be associated with participation. It is important to gain insight into QoL, patients' ability to perform their work, diet and dental consequences in long-term follow-up of HNC patients, to allow for evidence-based decision-making regarding treatment options for HNC.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for HNC with curative intent
* Finished treatment at least six months ago in the University Hospital Maastricht, MAASTRO Clinic or the University Medical Centre Groningen

Exclusion Criteria:

* Unable to read Dutch
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for head and neck cancer more than 6 months ago.
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Maastricht Radiation Oncology, Maastricht, Limburg
  - University Medical Center Groningen, Department of Radiation Oncology, Groningen, Provincie Groningen